CLINICAL TRIAL: NCT03047317
Title: A Phase I Pharmacokinetic Study of MABp1 in Healthy Volunteers
Brief Title: A Pharmacokinetic Study of MABp1 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-PT041
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MABp1 (Experimental)
  Interventions: Biological: MABp1

INTERVENTIONS:
Biological: MABp1 — Single dose of intravenous MABp1

SUMMARY:
This is an open label study of MABp1 in six healthy volunteers. Participants will receive a single infusion of MABp1 at the 7.5 mg/kg IV dose. Participants will undergo blood sampling for pK analysis at 15 times points during the course of 2 weeks (pre-infusion, 0.5 hr, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 5 hr, 6 hr, 12 hr, 24 hr, 48 hr, 96 hr, 192 hr, and 336 hr). In addition to pharmacokinetic data, participants will be monitored for the development of treatment emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18
2. Adequate bone marrow function as defined as:

   * absolute neutrophil count (neutrophil and bands) of ≥ 1,500/mm3 (≥ 1.5 x 109/L)
   * platelet count > 150,000/mm3
   * hemoglobin of ≥ 10 g/dL
3. Adequate renal function, defined by serum creatinine ≤ 1.5 x lab ULN.
4. Adequate hepatic function defined as:

   * total bilirubin ≤ 1.5 times lab ULN.
   * alanine aminotransferase (ALT) ≤ 2.0 times lab ULN.
5. For WOCBP, a negative pregnancy test at screening. For subjects with reproductive potential, a willingness to utilize contraception during the study and for at least 3 months after study completion. Sexually active men must use an accepted method of contraception during the study and for at least 3 months after study completion.
6. Signed and dated Institutional Review Board (IRB) approved informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

1. Treatment with any biologicals (including intravenous immunoglobulin) or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
2. Uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within the past 6 months.
   * Uncontrolled angina within the past 3 months.
   * Congestive heart failure within the past 3 months, defined as New York Heart Association (NYHA) Classes II or higher.
   * Uncontrolled hypertension (blood pressure >150 mm Hg systolic and >95 mm Hg diastolic).
3. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
4. Treatment with immunosuppressant agents, including corticosteroids or cyclosporine within the last 4 weeks.
5. Serious uncontrolled medical disorders, such as uncontrolled diabetes, active peptic ulcer disease, recent stroke (within 3 months), ongoing congestive heart failure, and any other condition, which in the opinion of the investigator, would put the subject at risk by participation in the protocol.
6. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
7. Infectious disease:

   * CRP >30 mg/L, or infection requiring treatment with antibiotics within 3 weeks prior to Screening,
   * Positive HIV, RPR, Hepatitis C antibody, or IGRA
8. Immunodeficiency by history.
9. Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding.
10. Major surgery within 28 days prior to Day 0.
11. WOCBP or men whose sexual partners are WOCBP who are unwilling or unable to use an acceptable method of contraception for at least 1 month prior to randomization, for the duration of the study, and for at least 3 months after the last dose of study medication.
12. History of progressive multifocal leukoencephalopathy or other demyelinating disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration | 2 weeks
  Pharmacokinetics--blood levels of MABp1 antibody
Time to Peak Plasma Concentration | 2 weeks
  Pharmacokinetics--blood levels of MABp1 antibody
Half Life | 2 weeks
  Pharmacokinetics--blood levels of MABp1 antibody
Area under the plasma concentration versus time curve | 2 weeks
  Pharmacokinetics--blood levels of MABp1 antibody

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events | 2 weeks
  The occurrence and incidence of treatment emergent adverse events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stecher, MD, Study Director — XBiotech, Inc.
Locations (1):
- XBiotech Investigative Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No